CLINICAL TRIAL: NCT03700242
Title: Imovax® Rabies and VERORAB® Immunogenicity and Safety After One Week 2-sites Intradermal or 1-site Intramuscular Pre-Exposure Prophylaxis Regimens, Followed by a Simulated Intradermal or Intramuscular Post-Exposure Prophylaxis Regimen at One Year
Brief Title: Imovax® Rabies and VERORAB® Immunogenicity and Safety After One Week 2-sites Intradermal or 1-site Intramuscular Pre-Exposure Prophylaxis Regimens, Followed by a Simulated Post-Exposure Prophylaxis Regimen at One Year
Acronym: VAJ00001
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAJ00001; U1111-1216-6210 (Other: UTN)
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Healthy Volunteers (Rabies Immunization)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Group 1 (Experimental): 1 IM dose of human diploid cell vaccine (HDCV) on D0 and D7 (short HDCV IM PrEP regimen), followed by 1 IM dose of HDCV on Year (Y)1 and Y1 + 3 days
  Interventions: Biological: HDCV
- Group 2 (Active Comparator): 1 IM dose of HDCV on D0, D7, and D21 (reference), followed by 1 IM dose of HDCV on Y1 and Y1 + 3 days
  Interventions: Biological: HDCV
- Group 3 (Experimental): 2 intradermal (ID) doses of HDCV on D0 and D7 (short HDCV ID PrEP regimen), followed by 1 ID dose of HDCV on Y1 and Y1 + 3 days
  Interventions: Biological: HDCV
- Group 4 (Experimental): 1 IM dose of purified Vero cell rabies vaccine (PVRV) on D0 and D7 (short PVRV IM PrEP regimen), followed by 1 IM dose of PVRV on Y1 and Y1 + 3 days
  Interventions: Biological: PVRV
- Group 5 (Experimental): 2 ID doses of PVRV on D0 and D7 (short PVRV ID PrEP regimen), followed by 1 ID dose of PVRV on Y1 and Y1 + 3 days
  Interventions: Biological: PVRV

INTERVENTIONS:
Biological: HDCV — Pharmaceutical form:Solution for injection Route of administration: Intramuscular
  Arms: Group 1; Group 2
Biological: HDCV — Pharmaceutical form:Solution for injection Route of administration: Intradermal
  Arms: Group 3
Biological: PVRV — Pharmaceutical form:Solution for injection Route of administration: Intramuscular
  Arms: Group 4
Biological: PVRV — Pharmaceutical form:Solution for injection Route of administration: Intradermal
  Arms: Group 5

SUMMARY:
The primary objective of the study is to demonstrate that a short intramuscular (IM) pre-exposure prophylaxis (PrEP) regimen is non-inferior to the reference IM PrEP regimen in terms of seroconversion rate.

The secondary objectives of the study are:

* To describe the immunogenicity of the PrEP regimen in each group
* To describe the antibody persistence in each group 6 months and 1 year after the last PrEP vaccination
* To describe the immunogenicity of the simulated post-exposure prophylaxis (PEP) regimen in each group
* To describe the safety profile of study vaccines administered as PrEP regimen and as a simulated PEP regimen in each group

DETAILED DESCRIPTION:
Study duration per participant is approximately 403 to 436 days

ELIGIBILITY:
Inclusion criteria :

* Aged ≥ 2 years on the day of inclusion
* Participant aged < 18 years: Assent form has been signed and dated by the subject (as appropriate, according to country-specific institution requirements), and informed consent form (ICF) signed and dated by the parent or another legally acceptable representative
* Participant aged ≥ 18 years: ICF signed and dated by the subject
* The participant (and parent/legally acceptable representative, if applicable) is able to attend all scheduled visits and to comply with all trial procedures

Exclusion criteria:

* Participant is pregnant, or lactating, or of childbearing potential and not using an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination until at least 4 weeks after the last vaccination. To be considered of non-childbearing potential, a female must be pre-menarche or post-menopausal for at least 1 year, or surgically sterile.
* Participation at the time of study enrollment (or in the 4 weeks preceding the first trial vaccination) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination or planned receipt of any vaccine in the 4 weeks following any trial vaccination except for influenza vaccination, which may be received at least 2 weeks before study vaccines. This exception includes monovalent pandemic influenza vaccines and multivalent influenza vaccines.
* Previous vaccination at any time against rabies with either the trial vaccine or another vaccine
* Receipt of immune globulins, blood, or blood-derived products in the past 3 months
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances
* Self-reported thrombocytopenia, contraindicating IM vaccination
* Bleeding disorder or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 38.0 C). A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study
* History of Guillain-Barré syndrome
* Receipt of chloroquine or other medications used for malaria chemoprophylaxis, with or without other anti-malarial treatment, for more than 4 weeks (duration of anti-malarial course) and part of the treatment received within the 2 weeks before vaccination, contraindicating intradermal vaccination

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 570 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2019-01-19 (Actual); Study Completion 2020-04-08 (Actual)

PRIMARY OUTCOMES:
Seroconversion of participant | 14 days after the last PrEP vaccination
  Rabies virus neutralizing antibodies (RVNA) titer ≥ 0.5 IU/mL

SECONDARY OUTCOMES:
Participant RVNA titer | Day 0 and 14 days after the last PrEP vaccination
Persistence of RVNA titer | 6 months and 1 year after the last PrEP vaccination
Participant RVNA titer after simulated PEP vaccination | 7 and 14 days after the first simulated PEP vaccination
Seroconversion of participant | Day 0 and 14 days after the last PrEP vaccination
  RVNA titer ≥ 0.5 IU/mL
Persistence of seroconversion | 6 months and 1 year after the last PrEP vaccination
  RVNA titer ≥ 0.5 IU/mL
Seroconversion of participant after simulated PEP vaccination - | 7 and 14 days after the first simulated PEPvaccination
  RVNA titer ≥ 0.5 IU/mL
Seropositivity of participant | Day 0 and 14 days after the last PrEP vaccination
  RVNA titer ≥ the lower limit of quantitation (LLOQ)
Persistence of seropositivity | 6 months and 1 year after the last PrEP vaccination
  RVNA titer ≥ the LLOQ
Seropositivity of participant after simulated PEP vaccination | 7 and 14 days after the first simulated PEP vaccination
  RVNA titer ≥ the LLOQ
Participant RVNA titer ratios | 14 days after last PrEP vaccination
  Titer 14 days after the last PrEP vaccination / titer at D0
Participant RVNA titer ratios (persistence assessment) | 6 months and 1 year after the last PrEP vaccination
  RVNA titer ratios are assessed 6 months / 14 days after the last PrEP vaccination, and 1 year / 14 days after the last PrEP vaccination
Participant RVNA titer after simulated PEP vaccination | 1 year after the last PrEP vaccination
  Ratio of titers measured 7 and 14 days after the first simulated PEP vaccination / 1 year after the last PrEP vaccination
Solicited injection site and systemic reactions after PrEP vaccination | 7 days after PrEP vaccination
  Injection site reactions: injection site pain, erythema, and swelling. Systemic reactions: fever, headache, malaise and myalgia.
Solicited injection site and systemic reactions after simulated PEP vaccination | 7 days after simulated PEP vaccination
  Injection site reactions: injection site pain, erythema, and swelling. Systemic reactions: fever, headache, malaise and myalgia. Solicited systemic reactions are collected between the first and second PEP injection and within 7 days after the second PEP injection.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (2):
- Philippines (2):
  - Investigational Site Number 002, Cebu City
  - Investigational Site Number 001, City of Muntinlupa

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Quiambao BP, Lim JG, Bosch Castells V, Augard C, Petit C, Bravo C, Delore V, Houillon G. One-week intramuscular or intradermal pre-exposure prophylaxis with human diploid cell vaccine or Vero cell rabies vaccine, followed by simulated post-exposure prophylaxis at one year: A phase III, open-label, randomized, controlled trial to assess immunogenicity and safety. Vaccine. 2022 Aug 26;40(36):5347-5355. doi: 10.1016/j.vaccine.2022.07.037. Epub 2022 Aug 3. PMID 35933278